CLINICAL TRIAL: NCT00381069
Title: Obesity Prevention and Control in Community Recreation Centers
Brief Title: SDSU MOVE/Me Muevo Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Elder, Albert W. Johnson Distinguished Professor Emeritus, Lecturer, San Diego State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DK72994; R01DK072994 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Childhood Obesity
Keywords: Recreation Centers; Families; Obesity Prevention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Family & Community Recreation Center Intervention — The two year intervention involves changing the environment and policies in community recreation centers to promote physical activity and healthy eating choices. The Recreation Specialist will meet with recreation center staff monthly to create action plans that work towards this goal. Family Health Coaches will be in contact with intervention families twice a month either through a phone consultation, workshop at the recreation center,or home visit. Intervention families will receive a monthly mailing highlighting tips for healthy eating and physical activity. MOVE families will be encouraged to utilize the recreation center as a resource in supporting their child's physical activity and healthy eating behaviors.
  Other Names: MOVE/me Muevo Family Health Program

SUMMARY:
The purpose of this study is to design, implement, and evaluate a recreation site-based obesity prevention & control intervention for 7-9 year old children and their families by targeting physical activity and dietary behaviors.

DETAILED DESCRIPTION:
The primary aim is to evaluate the effectiveness of a multi-level intervention to prevent the onset of overweight and obesity in 7-9 year old children. The recreation center site intervention emphasizes changes in quantity and quality of physical activity and nutrition-related offerings within the centers. The home site intervention targets the home environment and household rule setting delivered via Family Health Coaches and tailored to the needs of the family. Five hundred forty one (541) families were recruited to participate in this project. Participants were selected in part based on residence in proximity to participating recreation centers. Eighteen (18) families living up to 3 miles from each of the 30 recreation centers involved in the project were be recruited to participate. For each family, one child was recruited between the ages of 5 and 8 years old and this child's primary caregiver was enrolled in the study. The study's primary outcome is Body Mass Index (kg/m2).

Comparisons: Control vs. Intervention

ELIGIBILITY:
Inclusion Criteria:

* Primary residence within 3 miles of recreation center
* Children ages 5-8 at baseline
* Commit to participate in study for 3 1/2 years
* Participating parent must be a legal guardian of the child
* Parent and child must be able to speak and read English or Spanish
* Willing to be randomly assigned to control or intervention

Exclusion Criteria:

* Child has a medical/health/psychological condition or is taking a medication that may impact the child's physical activity, diet or weight to confound BMI
* Parent or child is unable to read and speak English or Spanish
* Family plans to move during the next 3 1/2 years

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 541 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
BMI (height & weight) at baseline, 1 year of intervention, and post intervention | February 2010-August 2010

SECONDARY OUTCOMES:
Child physical activity measured by wearing the ActiGraph accelerometer in a subsample of 1/3 of participants from each center | February 2010-August 2010
Questionnaire to assess Parent-reported nutrition and eating behaviors,rules about physical activity & nutrition in the home, and physical activity & sedentary behavior at baseline, 2 years, 3 years. | February 2010-August 2010

CONTACTS AND LOCATIONS:
Overall Officials: John P Elder, PhD, MPH, Principal Investigator — San Diego State University Graduate School of Public Health
Locations (1):
- Sdsu Move, San Diego, California, United States